CLINICAL TRIAL: NCT03737123
Title: A Phase II Trial of Atezolizumab Plus Chemotherapy After Progression on PD-1 or PD-L1 Inhibitor in Cisplatin-ineligible Patients With Advanced Urothelial Carcinoma: HCRN GU17-295
Brief Title: Trial of Atezolizumab Plus Chemotherapy After Progression on PD-1 or PD-L1 in Cisplatin-ineligible Patients With Advanced Urothelial Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Nabil Adra (Other)
Collaborators: Genentech, Inc. (Industry); Indiana University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Nabil Adra, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GU17-295
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Carboplatin; Gemcitabine; atezolizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Chemotherapy and Atezolizumab (Experimental): Subjects that received a PD 1 or PD-L1 inhibitor with no prior platinum chemotherapy for metastatic disease will be treated with atezolizumab + carboplatin + gemcitabine on trial. Subjects that received sequential or concurrent PD1/PDL1 inhibitor and carboplatin-based regimen will be treated with atezolizumab + docetaxel on trial.
  Interventions: Drug: Carboplatin; Drug: Gemcitabine; Drug: Atezolizumab; Drug: Docetaxel

INTERVENTIONS:
Drug: Carboplatin — Carboplatin AUC 4 IV Day 1 of each 21 day cycle
  Other Names: paraplatin
Drug: Gemcitabine — Gemcitabine 1,000 mg/m2 IV Day 1 and Day 8 of each 21 day cycle
  Other Names: Gemzar
Drug: Atezolizumab — Atezolizumab 1,200 mg IV Day 1 of each 21 day cycle
  Other Names: Tecentriq
Drug: Docetaxel — Docetaxel 75 mg/m2 IV Day 1 of each 21 day Cycle.
  Other Names: Taxotere

SUMMARY:
This is a single arm phase II study assessing the activity of atezolizumab in combination with carboplatin + gemcitabine or docetaxel compared to historical controls of chemotherapy only in metastatic or recurrent urothelial carcinoma subjects. Subjects that received a PD 1 or PD-L1 inhibitor with no prior platinum chemotherapy for metastatic disease will be treated with atezolizumab + carboplatin + gemcitabine on trial. Subjects that received sequential or concurrent PD1/PDL1 inhibitor and carboplatin-based regimen will be treated with atezolizumab + docetaxel on trial.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0-2 within 28 days prior to registration.
* Histological or cytological confirmed metastatic or unresectable locally advanced urothelial carcinoma (primary tumor: renal pelvis, ureters, urinary bladder, or urethra).
* Patients with mixed histologies are eligible.
* Cisplatin ineligible at the time of diagnosis with metastatic urothelial carcinoma based on consensus definition with any of the following criteria: ECOG PS 2, creatinine clearance < 60mL/min, CTCAE v4 grade ≥ 2 hearing loss, CTCAE v4 grade ≥ 2 peripheral neuropathy, New York Heart Association (NYHA) class ≥ 3 heart failure.
* Measurable disease according to RECIST 1.1 within 28 days prior to registration.
* Must have had progressive metastatic disease after previous treatment with PD-1 or PD-L1 inhibitor (in the adjuvant or metastatic setting). Treatment regimen will be determined based on prior treatment:

  * PD1 or PDL1 inhibitor with no prior platinum chemotherapy for metastatic disease. These patients should be treated with atezolizumab + carboplatin + gemcitabine on trial.
  * Sequential or concurrent PD1/PDL1 inhibitor and carboplatin-based regimen. These patients should be treated with atezolizumab + docetaxel on trial.
* Most recent therapy does not have to have been a checkpoint inhibitor. Intercurrent treatment is acceptable if subjects meet all other inclusion criteria.
* A subject with prior brain metastasis may be considered if they have completed their treatment for brain metastasis at least 4 weeks prior to study registration, have been off of corticosteroids for ≥ 2 weeks, and are asymptomatic.
* Previous neoadjuvant or adjuvant chemotherapy that was completed 6 months prior to study enrollment is allowed.
* REQUIRED archival tumor tissue (prior to treatment with single agent PD-1 or PD-L1 inhibitor) must be identified prior to registration and obtained during the screening period. Confirmation of acquisition should occur prior to C1D1 treatment. Unavailability of tissue will render the subject ineligible for study. Biopsy should be excisional, incisional or core needle. Fine needle aspiration is insufficient. Sample requirement is FFPE block + 1 H&E stained slide or 25 unstained slides + 1 H&E stained slide.
* Demonstrate adequate organ function as defined in the table below. All screening labs to be obtained within 28 days prior to registration.

  * White blood cell (WBC) ≥ 2 k/mm3
  * Absolute Neutrophil Count (ANC) ≥ 1.5 K/mm3
  * Hemoglobin (Hgb) ≥ 9 g/dL
  * Platelet >100k
  * Estimated creatinine clearance ≥ 30 mL/min
  * Bilirubin 1.5 ≤ (ULN)
  * Aspartate aminotransferase (AST) ≤ 1.5 × ULN
  * Alanine aminotransferase (ALT) ≤ 1.5 × ULN
  * International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤ 2 × ULN (Note: This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose)
* Females of childbearing potential (FOCBP) must have a negative serum pregnancy test within 28 days prior to registration. These women must also have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of atezolizumab then every 6 weeks thereafter. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is post-menopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 62 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL.
* Females of childbearing potential and males must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 150 days (5 months) after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method.
* Men who are sexually active with FOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving atezolizumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 150 days (5 months) after the last dose of investigational product.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

* Previous autoimmune complication from PD-1 or PD-L1 inhibitor requiring permanent discontinuation of therapy.
* Previous permanent discontinuation from PD-1 or PD-L1 inhibitor due to an adverse event (patients who had temporary holds or discontinuation of PD-1 or PD-L1 inhibitor and then re-treated are eligible).
* Any serious or uncontrolled medical disorder or active infection that would impair the ability of the subject to receive protocol therapy.
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* 5. Has a known additional malignancy that is progressing or required treatment ≤ 48 months of study registration. Exceptions: include malignancies with negligible risk of metastasis or death treated with expected curative outcome or undergoing surveillance per investigator's discretion (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, ductal carcinoma in situ treated surgically with curative intent, or very low risk or low risk prostate cancer per NCCN guidelines).
* Active central nervous system (CNS) metastases. Subjects with brain metastases are eligible if metastases have been treated and there is no magnetic resonance imaging (MRI) evidence of progression within 28 days prior to the first dose of atezolizumab administration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
* Treatment with any investigational drug within 30 days prior to registration.
* Subjects with an active or recent history of a known or suspected autoimmune disease or recent history of a syndrome that required systemic corticosteroids/immunosuppressive medications EXCEPT for syndromes which would not be expected to recur in the absence of an external trigger. (Subjects with vitiligo, autoimmune thyroiditis, or type I diabetes mellitus are permitted to enroll.).
* As there is potential for hepatic toxicity with atezolizumab, drugs with a predisposition to hepatoxicity should be used with caution in subjects treated with atezolizumab-containing regimen.
* Subjects should be excluded if they have known history of testing positive for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection. Testing is not required.
* Subjects should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). Testing is not required.
* History of allergy to atezolizumab or respective chemotherapy regimen (carboplatin + gemcitabine or docetaxel).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Adra, MD, Principal Investigator — Indiana University Melvin and Bren Simon Cancer Center
Locations (4):
- United States (4):
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Nebraska Methodist Hosptial, Omaha, Nebraska
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase IIA : Atezolizumab + Carboplatin + Gemcitabine: Subjects that received a PD 1 or PD-L1 inhibitor with no prior platinum chemotherapy for metastatic disease will be treated with atezolizumab + carboplatin + gemcitabine on trial.
  Carboplatin: Carboplatin AUC 4 IV Day 1 of each 21 day cycle
  Gemcitabine: Gemcitabine 1,000 mg/m2 IV Day 1 and Day 8 of each 21 day cycle
  Atezolizumab: Atezolizumab 1,200 mg IV Day 1 of each 21 day cycle
- Phase IIB : Docetaxel + Atezolizumab: Subjects that received sequential or concurrent PD1/PDL1 inhibitor and carboplatin-based regimen will be treated with docetaxel + atezolizumab on trial.
  Docetaxel: Docetaxel 75 mg/m2 IV Day 1 of each 21 day Cycle.
  Atezolizumab: Atezolizumab 1,200 mg IV Day 1 of each 21 day cycle.
Period: Study Treatment
Arm/Group | Phase IIA : Atezolizumab + Carboplatin + Gemcitabine | Phase IIB : Docetaxel + Atezolizumab
Started | 6 | 0
Completed | 0 | 0
Not Completed | 6 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Disease Progression | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Follow up
Arm/Group | Phase IIA : Atezolizumab + Carboplatin + Gemcitabine | Phase IIB : Docetaxel + Atezolizumab
Started (Treatment and Follow up both are at different time period. Therefore, the number of subjects to start follow up is not equal to the number of subjects who have completed treatment.) | 6 | 0
Completed | 0 | 0
Not Completed | 6 | 0
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Termination of study | 4 | 0

BASELINE CHARACTERISTICS:
Population: No subject had been enrolled in arm B of Phase II
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase IIA : Atezolizumab + Carboplatin + Gemcitabine | Phase IIB : Docetaxel + Atezolizumab | Total
Number analyzed (Participants) | 6 | 0 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 6 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 5 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 0 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG PERFORMANCE STATUS:
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 4 | 0 | 4
    1 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Evaluate PFS among patients to be treated with atezolizumab in combination with carboplatin + gemcitabine or docetaxel, who have cisplatin-ineligible metastatic urothelial carcinoma and who have progressed on prior PD-1 or PD-L1 inhibitor. PFS defined as duration from date of treatment start until progression according to RECIST 1.1 criteria, or death from any cause.
  Per RECIST 1.1 criteria, Progressive disease can be defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: From C1D1 until progression or death or up to a maximum of 26 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase IIA : Atezolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 6
months | 11.3 [3.2 to NA] — insufficient number of participants with events

2. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability of Carboplatin + Gemcitabine or Docetaxel
Description: Assess the safety and tolerability of the combination of atezolizumab plus chemotherapy (carboplatin + gemcitabine or docetaxel) using CTCAE v4.03. Number of subjects who had any adverse events or events greater than grade 3 were reported in this outcome measure.
Time Frame: From C1D1 until death or up to a maximum of 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase IIA : Atezolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 6
Participants
  Number of patients had at least one adverse event of any grade | 6
  Number of patients had at least one grade 3 or greater adverse event | 6
  Number of patients had at least one grade 3 or greater treatment related adverse event | 6
  Number of patients having serious adverse event | 3

3. Secondary Outcome: Objective Response Rate (ORR) With RECIST 1.1
Description: Objective response rate (ORR) using RECIST 1.1 defined as the proportion of all subjects with confirmed PR or CR according to RECIST 1.1, from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the start of treatment).
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: From C1D1 until death or up to a maximum of 28 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase IIA : Atezolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 5
percentage of participants | 40 [5.3 to 85.3]

4. Secondary Outcome: Objective Response Rate (ORR) With irRECIST
Description: ORR defined as the proportion of all subjects with confirmed PR or CR using immunerelated response criteria (irRECIST), from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the start of treatment).
  Per irRECIST for target lesions Complete Response (irCR), Disappearance of all target lesions; Partial Response (irPR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = irCR + irPR.
Time Frame: From C1D1 until death or up to a maximum of 28 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase IIA : Atezolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 5
percentage of participants | 40 [5.3 to 85.3]

5. Secondary Outcome: Clinical Benefit Rate (CBR) With RECIST 1.1
Description: Clinical benefit rate (CBR) of treatment (defined by proportion of all subjects with stable disease for at least 3 months, partial response, or complete response) using RECIST 1.1 from the start of treatment until disease/recurrence(taking as reference for progressive disease the smallest measurements recorded since the start of treatment). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions, neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter since the treatment started; Clinical Benefit Rate (CBR) = CR +PR +SD (for atleast 3 months).
Time Frame: From C1D1 until death or up to a maximum of 28 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase IIA : Atezolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 6
percentage of participants | 100 [47.8 to 100.0]

6. Secondary Outcome: Clinical Benefit Rate (CBR) With irRECIST
Description: Clinical benefit rate (CBR) of treatment (defined by proportion of all subjects with stable disease for at least 3 months, partial response, or complete response) using irRECIST from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the start of treatment).
  Per irRECIST for target lesions: Complete Response (irCR), Disappearance of all target lesions; Partial Response (irPR), >=30% decrease in the sum of the longest diameter of target lesions, neither sufficient shrinkage to qualify for irPR nor sufficient increase to qualify for irPD, taking as reference the smallest sum longest diameter since the treatment started; Clinical Benefit Rate (CBR) = irCR +irPR +irSD (for atleast 3 months).
Time Frame: From C1D1 until death or up to a maximum of 28 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase IIA : Atezolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 6
percentage of participants | 100 [47.8 to 100]

7. Secondary Outcome: PFS by irRECIST
Description: PFS defined as duration from date of treatment start until progression according to irRECIST criteria or death from any cause. Per irRECIST criteria, Progressive disease can be defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: From C1D1 until progression or death or up to a maximum of 26 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase IIA : Atezolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 6
months | 11.3 [5.3 to NA] — insufficient number of participants with events

8. Secondary Outcome: Overall Survival (OS)
Description: OS defined by the date of treatment start to date of death from any cause.
Time Frame: From C1D1 until death or up to a maximum of 28 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase IIA : Atezolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 6
months | NA [5.3 to NA] — insufficient number of participants with events

9. Secondary Outcome: Progression Free Survival (PFS) Compared to Historical Controls
Description: To compare Progression Free Survival(PFS) with the historical control, Null hypothesis - Patients receiving atezolizumab plus chemotherapy (carboplatin +gemcitabine or docetaxel) will have a median PFS of 4 months.
  Alternative hypothesis - Patients receiving atezolizumab plus chemotherapy (carboplatin + gemcitabine or docetaxel) will have a median PFS of 7.2 months.
  Progression Free Survival defined as duration from date of treatment start until progression according to RECIST 1.1 criteria, or death from any cause.Per RECIST 1.1 criteria, Progressive disease can be defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: From C1D1 until progression or death or up to a maximum of 26 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase IIA : Atezolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 5
months | 11.3 [3.2 to NA] — insufficient number of participants with events prevents determining the upper confidence interval

10. Secondary Outcome: Progression Free Survival (PFS) for Atezolizumab + Carboplatin and Gemcitabine
Description: Evaluate PFS for atezolizumab + carboplatin and gemcitabine. PFS defined as duration from date of treatment start until progression according to RECIST 1.1 criteria, or death from any cause.Per RECIST 1.1 criteria, Progressive disease can be defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: From C1D1 until death or progression or up to a maximum of 26 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase IIA : Atezolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 6
months | 11.3 [3.2 to NA] — insufficient number of participants with events

11. Secondary Outcome: Progression Free Survival (PFS) for Atezolizumab + Docetaxel
Description: Evaluate PFS for atezolizumab + docetaxel. PFS defined as duration from date of treatment start until progression according to RECIST 1.1 criteria, or death from any cause. Per RECIST 1.1 criteria, Progressive disease can be defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: From C1D1 until progression or death
Population: No subject was enrolled in this arm.
Arm/Group | Phase IIB : Docetaxel + Atezolizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From C1D1 for every treatment cycle of 21 days until death or up to a maximum of 8 months.
Description: No subjects had been enrolled in Phase II Arm B.
Arm/Group | Phase IIA : Atezolizumab + Carboplatin + Gemcitabine
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase IIA : Atezolizumab + Carboplatin + Gemcitabine (N=6)
ANEMIA (Blood and lymphatic system disorders) | 1 (1)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
STROKE (Nervous system disorders) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase IIA : Atezolizumab + Carboplatin + Gemcitabine (N=6)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (3)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 5 (29)
ANOREXIA (Metabolism and nutrition disorders) | 3 (4)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
CHEST PAIN - CARDIAC (Cardiac disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (2)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 3 (6)
DIZZINESS (Nervous system disorders) | 3 (6)
DUODENAL ULCER (Gastrointestinal disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 3 (9)
EDEMA LIMBS (General disorders) | 2 (3)
FALL (Injury, poisoning and procedural complications) | 1 (1)
FATIGUE (General disorders) | 3 (12)
FEVER (General disorders) | 2 (2)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1)
HEMATOMA (Vascular disorders) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 1 (2)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (3)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (2)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 1 (2)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 2 (2)
LIPASE INCREASED (Investigations) | 2 (4)
NAUSEA (Gastrointestinal disorders) | 3 (6)
NEUTROPHIL COUNT DECREASED (Investigations) | 3 (6)
PAIN (General disorders) | 3 (4)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (9)
PANCREATITIS (Gastrointestinal disorders) | 1 (1)
PARESTHESIA (Nervous system disorders) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 3 (4)
PLATELET COUNT DECREASED (Investigations) | 4 (10)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (3)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 2 (3)
SYNCOPE (Nervous system disorders) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 2 (2)
URINARY FREQUENCY (Renal and urinary disorders) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2)
URINARY TRACT PAIN (Renal and urinary disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
WEIGHT LOSS (Investigations) | 1 (1)
WHITE BLOOD CELL DECREASED (Investigations) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/23/NCT03737123/Prot_SAP_000.pdf